CLINICAL TRIAL: NCT01938768
Title: Effects of an Early Prehospital Administration of Tranexamic Acid on Hyperfibrinolysis in Multiple Trauma
Status: Completed | Type: Observational
Sponsor: University of Göttingen (Other)
Collaborators: Tem International GmbH, München, Germany (Unknown)
Responsible Party: Principal Investigator, Dr. med. Nils Kunze, Principal Investigator, University of Göttingen
Other Study IDs: ZARI-NK-2013-02
Record Dates: First submitted 2013-09-05; First posted 2013-09-10 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Hyperfibrinolysis; Haemorrhage; Mortality
Keywords: Multiple trauma; Polytrauma; Hyperfibrinolysis; Tranexamic acid; Thrombelastometry
MeSH Terms: conditions — Hemorrhage; Multiple Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Tranexamic acid: patients with multiple trauma who received tranexamic acid on the scene
- Non tranexamic acid: patients with multiple trauma who did not receive tranexamic acid on the scene

SUMMARY:
Severe external and internal bleedings are common in multiple trauma patients. Uncontrollable blood loss is the cause for about one third of all trauma deaths. A number of blood clotting mechanisms are known to be triggered by major blood losses. These mechanisms shall secure the organisms from loosing even more blood. To avoid an overshooting clotting behavior, inhibiting mechanisms occur as well. An important inhibiting (or fibrinolytic) mechanism is the fibrinolysis that is based on the conversion of plasminogen to plasmin. In severe bleeding situations this mechanism tends to overshoot and therewith contributes to the severity of the bleeding. This phenomena is called hyperfibrinolysis and is found in approximately one third of all multiple trauma patients. Mortality rates are increased in these patients. Tranexamic acid is an antifibrinolytic drug that inhibits the conversion from plasminogen to plasmin and therefore is able to limit the effects hyperfibrinolysis. A large study showed positive influence of tranexamic acid on mortality rates and blood loss in severely injured patients, when it was administered in an early clinical setting. In this study we want to answer the question wether a hyperfibrinolysis can be seen in an early prehospital (on the scene) setting and how it is influenced by an early prehospital administration of tranexamic acid.

DETAILED DESCRIPTION:
In patients suffering from multiple trauma the initially responding emergency physician on the scene will take a blood sample for thrombelastometry immediately after i.v. access is established. According to the initial trauma life support protocols a number of patients will receive a dose of tranexamic acid during the initial treatment on the scene or during transport to the hospital. A second blood sample will be taken after arrival in the resuscitation area of the hospital. Thrombelastometric measurements will be performed with both blood samples and the extent of hyperfibrinolysis in both samples will be compared. In a second step the outcome of the patients who received tranexamic acid on the scene will be compared to those who did not receive the drug before reaching hospital.

ELIGIBILITY:
Inclusion Criteria:

* Multiple trauma ISS > 15
* Age > 18 years

Exclusion Criteria:

* No informed consent
* Inclusion to an interventional clinical trial
* Death of the patient on the scene or before the hospital was reached
* Delayed thrombelastometric measurement (> 4 hours)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited by emergency physicians on the scene by taking a blood sample for thrombelastometry.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2013-11; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Initial state of hyperfibrinolysis | Minutes after arrival on the scene
  State of hyperfibrinolysis quantified by thromelastometry and PAP-Complex (Plasmin-Antiplasmin-Complex) from a blood sample taken a soon as possible on the scene
State of hyperfibrinolysis on hospital admission | minutes to hours after incident
  State of hyperfibrinolysis quantified by thrombelastometry and PAP-Complex from a blood sample taken as soon as possible after hospital arrival

SECONDARY OUTCOMES:
transfusion of packed red blood cells | 48 hours
  units of packed RBC units transfused within 48 hours after hospital admission
substitution of coagulation products | 48 hours after hospital admission
  number and type of coagulation products given within 48 hours after hospital admission
length of stay intensive care unit (LOS ICU) | one year
  length of the first ICU stay
length of hospital stay | one year
  length of stay in the acute care hospital (not rehabilitation facilities)
mortality | 90 days
  dead within 90 days after hospital admission

CONTACTS AND LOCATIONS:
Overall Officials: Quintel Michael, Prof. Dr., Study Chair — University of Goettingen; Roessler Markus, PD Dr., Study Director — University of Goettingen
Locations (1):
- University Medical Center Göttingen, Göttingen, Lower Saxony, Germany

REFERENCES:
- [Background] Schochl H, Frietsch T, Pavelka M, Jambor C. Hyperfibrinolysis after major trauma: differential diagnosis of lysis patterns and prognostic value of thrombelastometry. J Trauma. 2009 Jul;67(1):125-31. doi: 10.1097/TA.0b013e31818b2483. PMID 19590321
- [Background] CRASH-2 trial collaborators; Shakur H, Roberts I, Bautista R, Caballero J, Coats T, Dewan Y, El-Sayed H, Gogichaishvili T, Gupta S, Herrera J, Hunt B, Iribhogbe P, Izurieta M, Khamis H, Komolafe E, Marrero MA, Mejia-Mantilla J, Miranda J, Morales C, Olaomi O, Olldashi F, Perel P, Peto R, Ramana PV, Ravi RR, Yutthakasemsunt S. Effects of tranexamic acid on death, vascular occlusive events, and blood transfusion in trauma patients with significant haemorrhage (CRASH-2): a randomised, placebo-controlled trial. Lancet. 2010 Jul 3;376(9734):23-32. doi: 10.1016/S0140-6736(10)60835-5. Epub 2010 Jun 14. PMID 20554319
- [Background] CRASH-2 collaborators; Roberts I, Shakur H, Afolabi A, Brohi K, Coats T, Dewan Y, Gando S, Guyatt G, Hunt BJ, Morales C, Perel P, Prieto-Merino D, Woolley T. The importance of early treatment with tranexamic acid in bleeding trauma patients: an exploratory analysis of the CRASH-2 randomised controlled trial. Lancet. 2011 Mar 26;377(9771):1096-101, 1101.e1-2. doi: 10.1016/S0140-6736(11)60278-X. PMID 21439633
- [Derived] Kunze-Szikszay N, Krack LA, Wildenauer P, Wand S, Heyne T, Walliser K, Spering C, Bauer M, Quintel M, Roessler M. The pre-hospital administration of tranexamic acid to patients with multiple injuries and its effects on rotational thrombelastometry: a prospective observational study in pre-hospital emergency medicine. Scand J Trauma Resusc Emerg Med. 2016 Oct 10;24(1):122. doi: 10.1186/s13049-016-0314-4. PMID 27724970